CLINICAL TRIAL: NCT01672255
Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, SSRI and Exercise
Brief Title: Hypoglycemia Associated Autonomic Failure in Type 1 Diabetes Mellitus (DM)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00044537; SSRI and Exercise
Record Dates: First submitted 2012-08-17; First posted 2012-08-24 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes; Hypoglycemia Associated Autonomic Failure
Keywords: exercise; diabetes; SSRIs
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Diabetes Mellitus | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Trial 1-SSRI (Active Comparator): 90 minute exercise baseline with 6 weeks treatment with SSRI (Prozac). Repeat 90 minute exercise after 6 week treatment.
  Interventions: Drug: Fluoxetine
- Trial 2-Placebo (Placebo Comparator): 90 minute exercise at baseline with 6 weeks treatment with placebo. Repeat 90 minute exercise after 6 weeks treatment of placebo.
  Interventions: Drug: Placebo control

INTERVENTIONS:
Drug: Fluoxetine — 20 mg week 1, 40 mg week 2, 60 mg week 3, 80 mg week 4-6
  Other Names: Prozac
  Arms: Trial 1-SSRI
Drug: Placebo control — 20 mg Week 1, 40 mg Week 2, 60 mg Week 3, 80 mg Week 4-6
  Arms: Trial 2-Placebo

SUMMARY:
Exercise is a cornerstone of diabetes management. It helps reduce blood pressure, promote weight loss, lower insulin resistance and improve glucose and lipid (triglyceride and HDL-cholesterol) profiles. Unfortunately, the benefits of exercise are often not embraced by diabetic individuals because of the fear of low blood sugar (hypoglycemia). My laboratory has demonstrated that Autonomic nervous system (ANS) counterregulatory failure plays an important role in exercise associated hypoglycemia in Type 1 DM. ANS responses are significantly reduced in Type 1 DM and are further blunted by antecedent episodes of hypoglycemia. Furthermore, there is a large sexual dimorphism of reduced ANS responses during submaximal exercise in both Type 1 DM and healthy individuals that is unexplained. Accumulating data are demonstrating that serotonergic pathways can regulate ANS discharge. Generally, serotonergic pathways are inhibitory but both single and longer term administration of selective serotonin reuptake inhibitors (SSRI's) such as Prozac has been demonstrated to increase basal epinephrine levels and enhance baroreflex control of Sympathetic nervous system (SNS) activity. What is unknown is whether fluoxetine can also enhance SNS responses and also override the large ANS sexual dimorphism present during sub maximal exercise. Therefore, the purpose of this study is to determine if the SSRI fluoxetine (Prozac) can improve SNS responses during exercise.

ELIGIBILITY:
Inclusion Criteria:

* 32 (16 males, 16 females) Healthy controls aged 18-45 yr.
* 32 (16 males, 16 females) Type 1 diabetic patients aged 18-45 yr.
* HbA1c 6-10.0%
* Has been diagnosed Type 1 DM
* No clinically diagnosed diabetic tissue complications (i.e. history of retinopathy, neuropathy, stasis ulcers, etc)
* Body mass index < 40kg • m-2

Exclusion Criteria:

* Pregnant women
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs, anemic or with known bleeding diatheses
* Subjects taking any of the following medications will be excluded: Non-selective Beta Blockers, Sedative-Hypnotics, Anticonvulsants, Antiparkinsonian drugs, Antipsychotics, Antidepressants, Mood stabilizers, CNS Stimulants, Opioids, Hallucinogens
* Subjects with a recent medical illness
* Subjects with a history of hypertension, heart disease, cerebrovascular incidents
* Current tobacco use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2012-10; Primary Completion 2025-05 (Actual); Study Completion 2025-05 (Actual)

PRIMARY OUTCOMES:
Change in Catecholamines | During 90 minute experimental period
  This change in catecholamines will be compared to another 90 minute experimental period after 8 weeks administration of SSRI or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MBBS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No